CLINICAL TRIAL: NCT05896072
Title: Comparison of the Effects of Ultrasound-Guided Erector Spinae Plane Block and Caudal Block on Postoperative Pain in Children Undergoing Unilateral Inguinal Hernia Operation
Brief Title: Comparison of Two Different Analgesic Regional Block Techniques in Pediatric Patients Undergoing a Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Abant Izzet Baysal University (Other)
Collaborators: Karabuk University (Other); Başakşehir Çam & Sakura City Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AIBU-TF-AR-II-003
Record Dates: First submitted 2023-05-04; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-06

CONDITIONS: Post Operative Pain; Inguinal Hernia
Keywords: Caudal block; Erector spinae block; Pediatric postoperative analgesia; Inguinal hernia
MeSH Terms: conditions — Pain, Postoperative; Hernia, Inguinal

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ESP Group (Experimental): Erector Spinae Plane Block Group
  Drug: 0,25% Bupivacaine 0,5ml/kg (max.20ml) will be used for blocks
  Interventions: Procedure: Erector Spinae Plane Block
- Caudal Group (Active Comparator): Caudal Block Group
  Drug: 0,25% Bupivacaine 0,5ml/kg (max.20ml) will be used for blocks
  Interventions: Procedure: Caudal Block

INTERVENTIONS:
Procedure: Erector Spinae Plane Block — Application of ultrasound-guided erector spinae plane block for perioperative analgesia for elective inguinal hernia repair. Erector spinae plane block will be administered under general anesthesia before the surgery
  Drug: Bupivacaine (Block Drug)
  For block performances, 0,25% Bupivacaine will be used at 0,5 ml/kg (max. 20cc).
  Arms: ESP Group
Procedure: Caudal Block — Application of caudal block for perioperative analgesia for elective inguinal hernia repair. The caudal block will be administered under general anesthesia before the surgery.
  Drug: Bupivacaine (Block Drug)
  0,25% Bupivacaine will be used at 0,5 ml/kg (max. 20cc) for block performances
  Other Names: Caudal Epidural Block
  Arms: Caudal Group

SUMMARY:
Lower abdominal operations; especially inguinal hernia repairs are one of the most frequently performed operations in the daily practice of pediatric surgeries.Regional anesthesia techniques are frequently and effectively used methods in postoperative pain control. Main purpose of this study is to compare the analgesic effect of ultrasound-guided erector spinae plane block and caudal block in pediatric unilateral inguinal hernia operations

DETAILED DESCRIPTION:
Patient mobilization and providing adequate analgesia are important components of perioperative care in the day case procedures.Providing adequate postoperative analgesia in the pediatric age group is also important in terms of future pain perception and the development of chronic pain in the next period. Regional anesthesia techniques are very effective and frequently used methods in pain control in children.While central blocks such as caudal epidural block, spinal block are frequently used in inguinal surgeries in children, they have been used in peripheral blocks and successful results have been obtained. Although central blocks are frequently used in the pediatric population, depending on the relevant surgical site, due to the difficulty of application and the capacity to create motor block, the peripheral blocks are among the alternative methods. Although ESP (Erector spinae plane) block is an interfascial plane block, anatomical studies support the idea that some of its clinical benefit may be due to its extension into the paravertebral and epidural space. Its use for pediatric abdominal surgeries has also been reported. Simple randomization will be used in randomization. With 5% margin of error, 80% Power, the standard effect size was determined as 0,72. Pediatric patients in the ASA I-II group, aged 1-8 years, who will undergo elective unilateral inguinal hernia operation under general anesthesia, will be sufficient to include n= 30 cases in each group.The investigators plan to conduct a prospective randomized controlled study for pediatric day case inguinal hernia surgeries. Oral midazolam (0.5 mg/kg) will be given to all children as premedication. After standard monitoring with pulse oximetry, electrocardiography and noninvasive blood pressure measurement in the operating room, anesthesia will be induced with air in 8% sevoflurane and 50% oxygen. Then, a 24-gauge intravenous (iv) cannula will be placed and 1 µg/kg fentanyl and 2-3 mg/kg propofol will be administered for anesthesia induction. The airway will be secured with the ProSeal laryngeal mask airway (Intravent-Orthofix, Maidenhead, UK). Anesthesia will be maintained with 50% nitrous oxide and 2% sevoflurane in oxygen. Additional opioid medication use during the operations will be recorded. At the end of the surgery, all patients will be given acetaminophen 10 mg/kg iv for postoperative analgesia. All blocks will be done after the airway is secured before the surgery begins. Patients will be placed in the side-lying position for ESP block. Following skin preparation with 10% povidone iodine, the ultrasound probe will be placed 1-2 cm lateral to the midline at the sacral level. L1 level will be determined by counting upwards from the sacrum. After identification of the erector spinae muscle (ESM) and the transverse process, a block needle will be inserted deep into the ESM in the cranio-caudal direction using an in-plane technique. Correct needle position will be confirmed by the application of 0.5-1 ml local anesthetic (LA). For block efficacy a pre-calculated dose (0.5 ml/kg) of 0.25% bupivacaine (maximum dose is limited to 20 ml) will be used. In the caudal group the patients will be placed in the side-lying position for the caudal block. The sacral cornues will be palpated and the block needle will be advanced at an angle of 45 degrees.After the needle hits the sacrum the angle will be reduced and retract few millimeters in the epidural space in the sacral canal. It will be checked that there is no blood and cerebrospinal fluid with negative aspiration. Bupivacaine will be administered at the same dose, at a dose of %0.25, 0.5 ml/kg (the maximum dose is limited to 20 ml). A pain nurse was scheduled to assess pain using the Face, Legs, Activity, Crying, and Consolability (FLACC) scores both in the postoperative recovery room and in the ward. FLACC scores will be recorded at 0, 1, 2, 4, 6, 12, and 24 hours postoperatively. Additional analgesia was planned according to the FLACC scores of the patients. If the FLACC score is between 2 and 4, acetaminophen 10 mg/kg iv was planned as additional analgesia in the ward, and tramadol 1 mg/kg iv was planned as an additional analgesic if the FLACC score was > 4. Patients can be discharged after 6 hours postoperatively. Parents will be informed about pain assessment and instructed to give 10 mg/kg oral acetaminophen if FLACC scores are between 2 and 4, and 7 mg/kg oral ibuprofen if FLACC scores are 4 or more. Analgesic requirements in the first 24 hours postoperatively, time to first analgesia, and parental satisfaction with analgesia provided will be recorded at postoperative follow-up visits by one of the anesthetists who are unfamiliar with the study groups. Parental satisfaction levels will be recorded as a numerical scale from 1 to 10; 1 will represent the lowest possible satisfaction level and 10 the highest satisfaction level.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patient scheduled for unilateral elective inguinal hernia operation
* ASA status 1-2

Exclusion Criteria:

* Pediatric patient's parents refusal
* Contraindications to regional anesthesia
* Known allergy to local anesthetics,
* Bleeding diathesis,
* Severe kidney or liver disease
* Presence of infection at the needle entry site.

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Estimated)
Dates: Start 2023-05-08 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Analgesic consumption | 24 Hour
  Opioid consumption, need for rescue analgesic

SECONDARY OUTCOMES:
The Face, Legs, Activity, Cry and Consolability (FLACC) scale for pediatric pain evaluation. | 24 Hour
  FLACC scale ( Face, legs, activity, cry and consolability scale) is an observational scale comprised five behavioural indicators that are scored from zero to two. The pain score is the sum of the item scores and ranges from zero to 10.Pain severity will be assessed on the FLACC scale from 0 to 10. A score of zero will be considered no pain and a score of 10 will be considered the most severe pain.
Parental Satisfaction Assessment | 24 Hour
  Satisfaction level of parents after pediatric will be saved as a numerical scale from 1 to 10; 1 will represent the lowest possible satisfaction level and 10 the highest satisfaction level.

CONTACTS AND LOCATIONS:
Overall Officials: Kenan Kart, MD, Principal Investigator — Karabuk University Training and Research Hospital; Kasım İlker İtal, Study Director — Bolu Abant University Hospital; Duygu Taskin, Study Chair — Karabuk University Training and Research Hospital
Locations (6):
- Turkey (Türkiye) (6):
  - Abant İzzet Baysal Education and Training Hospital, Bolu, Merkez
  - Bolu Abant İzzet Baysal Medical School, Bolu
  - Bolu Abant İzzet Baysal University Faculty of Medicine, Bolu
  - Karabuk University Karabuk Training and Research Hospital, Karabük
  - Karabuk University Training and Research Hospital, Karabük
  - Karabük University Training and Research Hospital, Karabük

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Result] Aksu C, Sen MC, Akay MA, Baydemir C, Gurkan Y. Erector Spinae Plane Block vs Quadratus Lumborum Block for pediatric lower abdominal surgery: A double blinded, prospective, and randomized trial. J Clin Anesth. 2019 Nov;57:24-28. doi: 10.1016/j.jclinane.2019.03.006. Epub 2019 Mar 6. PMID 30851499
- [Result] Cosarcan SK, Mahli A. [Comparison of intraoperative and postoperative analgesic properties of ilioinguinal/iliohypogastric and sacral epidural block in pediatric unilateral inguinal hernia operations]. Agri. 2022 Jan;34(1):38-46. doi: 10.14744/agri.2021.48254. Turkish. PMID 34988963